CLINICAL TRIAL: NCT03954197
Title: Evaluation of Priming Before in Vitro Maturation for Fertility Preservation in Breast Cancer Patients: a Randomized Controlled Study
Brief Title: Evaluation of Priming Before in Vitro Maturation for Fertility Preservation in Breast Cancer Patients
Acronym: PRIMIV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hôpital Jean Verdier (Other)
Responsible Party: Principal Investigator, Michael Grynberg, Professor, Hôpital Jean Verdier
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2014-A00819-38
Record Dates: First submitted 2019-05-16; First posted 2019-05-17 (Actual); Last update posted 2019-05-20 (Actual); Status verified 2019-05

CONDITIONS: Fertility Preservation; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — ricin A-GnRH conjugate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Without injection group (Experimental): no injection used as priming
  Interventions: Other: hCG; Other: GnRH a
- hCG group (Active Comparator): hCG used as priming
  Interventions: Other: No hormone; Other: GnRH a
- GnRHa group (Active Comparator): GnRH agonist used as priming
  Interventions: Other: No hormone; Other: hCG

INTERVENTIONS:
Other: No hormone — No hormonal injection before oocytes retrieval
  Arms: GnRHa group; hCG group
Other: hCG — a subcutaneous injection of hCG (Choriogonadotropin alpha, Ovitrelle®, Merck Serono, 250 µg) is performed 36 hours before oocytes retrieval
  Arms: GnRHa group; Without injection group
Other: GnRH a — a subcutaneous injection of GnRH agonist (triptorelin, Decapeptyl, Ipsen, 0,2 mg) is performed 36 hours before oocytes retrieval
  Arms: Without injection group; hCG group

SUMMARY:
Oocyte vitrification after in vitro maturation (IVM) is one of the main techniques for preserving female fertility before chemotherapy for breast cancer. In this technique, originally developed for patients with ovarian pathology, polycystic ovarian syndrome, induction of an LH peak has been shown to improve outcomes. Young women with breast cancer, who are candidates for urgent fertility preservation, do not have ovarian pathology. The objective of the present study is to assess whether the absence of therapeutic intervention prior to oocyte retrieval for IVM in these patients is at least as effective as the injection of hCG or GnRH agonist used in routine practice.

DETAILED DESCRIPTION:
In vitro maturation (IVM) is an assisted reproductive technology which consists in the retrieval of immature cumulus-oocyte complexes (COCs) from small antral follicles, followed by their in vitro maturation in specific culture conditions. Oocytes having reached metaphase II (MII) stage after 24 to 48 hours of IVM can then be fertilized. This procedure was first developed for patients presenting polycystic ovarian syndrome (PCOS), in order to avoid ovarian hyperstimulation syndrome (OHSS), an iatrogenic consequence of exogenous gonadotropins administration. However, the increasing use of GnRH antagonist protocols allowing ovulation trigger with GnRH agonist has dramatically reduced the indication of IVM in women at risk of OHSS. Yet, evidence indicate that IVM may be considered for patients presenting FSH resistance or contraindications to controlled ovarian stimulation. The recent development of female fertility preservation (FP) renewed interest to this technique. Indeed, it can be performed without any prior ovarian stimulation and whatever the phase of the menstrual cycle. Although it is still considered experimental, oocyte vitrification following IVM has been applied in different groups of patients, in particular those diagnosed with breast cancer, autoimmune or ovarian diseases. In physiologic conditions, final follicular maturation is induced by a double FSH and LH release which occurs when the dominant follicle reaches approximately 17 to 20 mm in diameter. This gonadotropin surge usually precedes the follicular rupture and mature oocyte release from 36 to 40 hours. In case of an assisted reproductive treatment, two strategies can be used to reproduce this hormonal signal: (i) either an injection of hCG, which binds to the LH receptor on granulosa cells, (ii) or a GnRH agonist (GnRHa) administration which induces an endogenous double peak of LH and FSH through a "flare up effect". Miming common practice for in vitro fertilization, priming with hCG or GnRHa injection 36 hours before the COCs retrieval has been suggested for patients undergoing IVM procedure in order to improve oocyte maturation rates and further IVM outcomes. Indeed, it is hypothesized that these iatrogenic hormonal activities might enhance the final oocyte maturation in vivo, therefore shortening the duration of the overall IVM process. Actually, in PCOS patients, several line of evidence indicate that IVM outcomes are improved after hCG priming. This positive effect might be explained by a premature expression of LH receptors on granulosa cells of small antral follicles <10 mm in diameter. Nevertheless, in normo-ovulatory non PCOS patients, LH receptor expression in these follicles remains very low, questioning the relevance of providing LH activity to improve oocyte maturation during IVM cycles performed for FP. The present investigation aimed to test whether the absence of therapeutic intervention prior to oocyte retrieval modifies IVM outcomes when compared with cycles primed either with recombinant hCG or GnRH agonist in breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 38 years;
* diagnosis of breast cancer (BC)
* indication for neoadjuvant chemotherapy;
* body mass index (BMI) ≤27kg/m2; regular ovulatory cycles;
* transvaginal ultrasound showing the presence of two ovaries with an antral follicle count (AFC) between 10 and 30 follicles;
* affiliation to the national social security system.
* Written informed consent was obtained from all participants

Exclusion Criteria:

* - previous chemotherapy, ovarian surgery or endometrioma;

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 204 (Estimated)
Dates: Start 2014-09-09 (Actual); Primary Completion 2019-09-09 (Estimated); Study Completion 2019-10-09 (Estimated)

PRIMARY OUTCOMES:
total number of mature oocytes cryopreserved | 4 days
  Total number of mature oocytes obtained and cryopreserved after IVM

SECONDARY OUTCOMES:
number of COCS recovered | 36 hours
  Total number of COCs recovered after COCs retrieval
maturation rate | 4 days
  ratio between the number of mature oocytes over the number of COCs recovered

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Jean Verdier, Bondy, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sonigo C, Le Conte G, Boubaya M, Ohanyan H, Presse M, El Hachem H, Cedrin-Durnerin I, Benoit A, Sifer C, Sermondade N, Grynberg M. Priming Before In Vitro Maturation Cycles in Cancer Patients Undergoing Urgent Fertility Preservation: a Randomized Controlled Study. Reprod Sci. 2020 Dec;27(12):2247-2256. doi: 10.1007/s43032-020-00244-0. Epub 2020 Jul 2. PMID 32617881